CLINICAL TRIAL: NCT03348618
Title: A Multi-site, Open-Label, Pilot Study to Evaluate the Benefit of Octagam 5%® in Subjects With Pediatric Acute-onset Neuropsychiatric Syndrome (PANS)
Brief Title: A Study to Evaluate the Benefit of Octagam 5%® in Subjects With Pediatric Acute-onset Neuropsychiatric Syndrome (PANS)
Acronym: PANS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IMMUNOe Research Centers (Industry)
Collaborators: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIS201701-PANS
Record Dates: First submitted 2017-11-14; First posted 2017-11-21 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-03

CONDITIONS: Pediatric Acute-Onset Neuropsychiatric Syndrome; Pediatric Autoimmune Neuropsychiatric Disorders Associated With Streptococcal Infections
Keywords: Obsessive-Compulsive Disorder; Anxiety; PANS; PANDAS; Children
MeSH Terms: conditions — Pediatric acute-onset neuropsychiatric syndrome; Pediatric Autoimmune Neuropsychiatric Disorders Associated with Streptococcal infections; Obsessive-Compulsive Disorder; Anxiety Disorders | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- IVIG (Experimental): IVIG dose at 1 g/Kg/body weight
  Interventions: Biological: IVIG

INTERVENTIONS:
Biological: IVIG — Intravenous immunoglobulin
  Other Names: Octagam 5%

SUMMARY:
This study will evaluate the use of intravenous immunoglobulins (IVIG) at a dose of 1g/Kg/body weight given every three weeks for 6 infusions in pediatric subjects ages 4 - 16 years with moderate to severe PANS. The study will compare biomarkers and behavioral scales before treatment, after the last infusion, 2 months, and at a minimum 6 months post-treatment.

DETAILED DESCRIPTION:
IVIG at an immunomodulatory dose of 1 g/Kg body weight has been known to induce suppression of systemic inflammation and has been used in the treatment of autoimmune diseases. It has been proven beneficial in inflammatory conditions affecting the nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children, 4-16 years of age
* Diagnosis of moderate to severe PANS based on accepted criteria
* Must be willing to follow study procedures and comply with wash-out period
* If using prophylactic antibiotics, must be on stable dose for 3 months

Exclusion Criteria:

* History of rheumatic fever, including Sydenham chorea (the neurologic manifestation)
* Previous IVIG therapy within the last 6 months
* Allergic reactions to blood products
* Patients who, in the investigator's opinion, might not be suitable for the trial.
* Steroid use

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Estimated)
Dates: Start 2017-11-24 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Change in Anxiety Disorders Interview Schedule for DSM-IV, Child, Parent Versions (ADIS) | Measurements at baseline, one week post treatment (19 weeks), and 6 + months post-treatment (43 + weeks)
  ADIS Child and Parent Interviews are designed to diagnose children with emotional disorder, where anxiety is a prominent component. Problem behaviors and diagnoses include school refusal behavior, separation anxiety, social phobia, specific phobia, panic disorder, agoraphobia, OCD and PTSD. Assessment of ADHD allows for differentiation of inattentive type, hyperactive-type, and combined type.
Change in Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) | Measurements at baseline, one week post treatment (19 weeks), and 6 + months post-treatment (43 + weeks)
  The scale is a clinician-rated, 10-item scale, each item rated from 0 (no symptoms) to 4 (extreme symptoms) (total range, 0 to 40), with separate subtotals for severity of obsessions and compulsions.
Change in Yale Global Tic Severity Scale (YGTSS) | Measurements at baseline, one week post treatment (19 weeks), and 6 + months post-treatment (43 + weeks)
  The CY-BOCS rating scale is designed to rate the severity and type of symptoms in patients with obsessive compulsive disorder (OCD). Ratings of the characteristics of obsessive or compulsive ideation and actions on a scale of 0 - 4, with 0 as none and 4 as extreme.
Change in Clinical Global Impressions (CGI) | Measurements at baseline, one week post treatment (19 weeks), and 6 + months post-treatment (43 + weeks)
  CGI is a 3-item observer-rated scale used to measure symptom severity, global improvement, and therapeutic response. Items 1 and 2 are rated on a 7-point scale; item 3 is rated from 0 to 4
Change in biomarkers levels | Measurements at baseline, one week post treatment (19 weeks), and 6 + months post-treatment (43 + weeks)
  Neuro-immune biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Melamed, MD, Principal Investigator — IMMUNOe Research Centers
Locations (3):
- United States (3):
  - IMMUNOe Research Centers, Centennial, Colorado
  - Midwest Pediatrics, Papillion, Nebraska
  - Allergy, Asthma & Immunology Relief Research Institute, Charlotte, North Carolina

REFERENCES:
- [Background] Swedo SE, Leckman JF Rose NR. From research subgroup to clinical syndrome: Modifying the PANDAS criteria to describe PANS (Pediatric Acute-onset Neuropsychiatric Syndrome). Pediatr Therapeut 2012, 2:2.
- [Background] Chang K, Frankovich J, Cooperstock M, Cunningham MW, Latimer ME, Murphy TK, Pasternack M, Thienemann M, Williams K, Walter J, Swedo SE; PANS Collaborative Consortium. Clinical evaluation of youth with pediatric acute-onset neuropsychiatric syndrome (PANS): recommendations from the 2013 PANS Consensus Conference. J Child Adolesc Psychopharmacol. 2015 Feb;25(1):3-13. doi: 10.1089/cap.2014.0084. Epub 2014 Oct 17. PMID 25325534
- [Background] Swedo SE, Leonard HL, Garvey M, Mittleman B, Allen AJ, Perlmutter S, Lougee L, Dow S, Zamkoff J, Dubbert BK. Pediatric autoimmune neuropsychiatric disorders associated with streptococcal infections: clinical description of the first 50 cases. Am J Psychiatry. 1998 Feb;155(2):264-71. doi: 10.1176/ajp.155.2.264. PMID 9464208
- [Derived] Melamed I, Kobayashi RH, O'Connor M, Kobayashi AL, Schechterman A, Heffron M, Canterberry S, Miranda H, Rashid N. Evaluation of Intravenous Immunoglobulin in Pediatric Acute-Onset Neuropsychiatric Syndrome. J Child Adolesc Psychopharmacol. 2021 Mar;31(2):118-128. doi: 10.1089/cap.2020.0100. Epub 2021 Feb 18. PMID 33601937